CLINICAL TRIAL: NCT04827784
Title: The Evaluation Of The Efficacy Of Auriculotemporal Nerve Block In Temporomandibular Disorders
Brief Title: Auriculotemporal Nerve Block in TMJ Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Aras Erdil, Oral and Maxillofacial Surgeon, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaU2
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Temporomandibular Joint Disorders; Arthralgia of TMJ
Keywords: Auriculotemporal nerve block; Temporomandibular disorders; Physiotherapy; Anesthesia; Local
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: Participants whose Temporomandibular disorders (TMD)-related complaints continued despite occlusal stabilization splint, NSAIDs and centrally acting muscle relaxant treatments were administered a total of 3 doses of Auriculotemporal Nerve Block (ATNB).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Auriculotemporal Nerve Block Administration (Experimental): A total of 3 doses of Auriculotemporal Nerve Block (ATNB) were administered to involved participants. Local anesthetic solutions containing Articaine Hydrochloride (80 mg / 2 ml) and epinephrine bitartrate (0.02 mg / 2 ml) were used for ATNB application. The injections were repeated on follow-up visits in the first and fourth weeks. The maximal mouth opening amounts, pain intensity values (via VAS scale), and self-reported outcomes were evaluated at the pre-injection, first week, fourth week, and sixth-month follow-up controls.
  Interventions: Procedure: local anaesthetic injection

INTERVENTIONS:
Procedure: local anaesthetic injection — The head and neck of the condyle were detected by palpating the pretragal area. Then, the needle was inserted anterior to the junction of the tragus and the lobule. After 0.5 ml the solution was subcutaneously infiltrated, the needle was protruded until it touched the neck of the condyle. Aspiration was performed to avoid intravenous injections, and the remaining solution was injected thereafter.

SUMMARY:
The retrospective study aimed to evaluate the efficacy of the Auriculotemporal Nerve Block (ATNB) in achieving unrestricted mouth opening amount and in reducing the pain scores in those patients diagnosed with disc displacement with (DDWR) and without reduction (DDWOR) according to the Diagnostic Criteria for Temporomandibular Disorders, who could not benefit from noninvasive methods but did not want further invasion.

DETAILED DESCRIPTION:
The records of 410 patients referred to the Department of Oral and Maxillofacial Surgery with TMD symptoms were reviewed to determine the treatment modalities used and their outcomes. The subjects were examined and diagnosed according to the Turkish translation version of The Diagnostic Criteria for Temporomandibular Disorders (DC/TMD-Axis 1 questionnaire and examination form). The pain intensity, maximal mouth opening (MMO) amounts, and self-reported outcome variables of twenty-two patients who underwent non-invasive therapies (occlusal stabilization splints, behavioral modifications, physical therapy, pharmacotherapy) but did not benefit from them and volunteered for the ATNB instead of invasive therapies (arthrocentesis, arthroscopy, and discectomy) were also evaluated. Prior to the ATNB, written informed consent was obtained from each participant. Also, each participant was warned about complications of the ATNB before the administration, such as hematoma at the injection site, positive aspiration, and temporary anesthesia of the facial nerve.

ELIGIBILITY:
Inclusion Criteria:

* Underwent non-invasive therapies (occlusal stabilization splints, behavioral modifications, physical therapy, pharmacotherapy) but did not benefit from them and volunteered for the ATNB instead of invasive therapies (arthrocentesis, arthroscopy, and discectomy).

Exclusion Criteria:

Patients with

* Symptoms of the diseases possibly related to TMD (e.g., fibromyalgia, hypothyroidism, scleroderma, rheumatoid arthritis)
* Orofacial disorders that might have been responsible for the TMD symptoms (e.g., neuralgia, migraine, myositis, trauma, neuropathic pain, infections)
* Complications due to ATNB (e.g., temporary facial nerve palsy, hematoma, positive aspiration)
* History of invasive therapies or TMJ surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Baseline Pain Intensity | At the initial visit before starting anesthetic administration.
  Pain intensity was measured using a 10-point Visual Analog Scale (VAS), in which 0 referred to 'no pain', 5 referred to 'moderate pain,' and 10 referred to 'excruciating pain'. The patients were asked to mark their pain intensities on VAS scale.
Post-injection Pain Intensity | At six months follow-up visit
  Pain intensity was measured using a 10-point Visual Analog Scale (VAS), in which 0 referred to 'no pain', 5 referred to 'moderate pain,' and 10 referred to 'excruciating pain'. The patients were asked to mark their pain intensities on VAS scale.
Change From Baseline Maximal Mouth Opening on Post-Injection Follow Up Visits | At the first week, fourth week and sixth month.
  All patients' maximal mouth opening were measured and recorded as the distance between upper and lower right central incisors.

SECONDARY OUTCOMES:
Overall Satisfaction With The Applied Treatment | At the six-month follow-up visit
  Patients were asked dichotomously to define the ATNB as successful/unsuccessful, according to their experience. The patients' responses were recorded individually.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet K. Tümer, AssocProfDr, Study Director — Alanya Alaaddin Keykubat University
Locations (1):
- Tokat Gaziosmanpasa University, Faculty of Dentistry, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data regarding participants were made available in the manuscript

REFERENCES:
- [Background] NASCIMENTO, Mirella Marques Mercês do, et al. Anesthetic blockage of the auriculotemporal nerve and its clinical implications. Odontologia Clínico-Científica (Online), 2011, 10.2: 143-146.
- [Background] Ayesh EE, Ernberg M, Svensson P. Effects of local anesthetics on somatosensory function in the temporomandibular joint area. Exp Brain Res. 2007 Jul;180(4):715-25. doi: 10.1007/s00221-007-0893-4. Epub 2007 Feb 15. PMID 17588187
- [Result] Nascimento MM, Vasconcelos BC, Porto GG, Ferdinanda G, Nogueira CM, Raimundo RD. Physical therapy and anesthetic blockage for treating temporomandibular disorders: a clinical trial. Med Oral Patol Oral Cir Bucal. 2013 Jan 1;18(1):e81-5. doi: 10.4317/medoral.17491. PMID 23229236